CLINICAL TRIAL: NCT00144872
Title: Evaluation of Lamotrigine in Subjects With Absence Seizures
Brief Title: LAMICTAL (Lamotrigine) For The Treatment Of Absence Seizures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAM100118
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Seizure, Absence
Keywords: Absence Seizures; EEG; LTG; Typical Absence Epilepsy; Epilepsy; LAMICTAL
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Lamotrigine

ARMS (1):
- Subjects receiving lamotrigine (Experimental): Eligible subjects will receive chewable dispersible tablets of lamotrigine with a starting dose of 0.3 milligrams per kilogram administered orally.
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine will be given as chewable dispersible tablets with dosing strengths of 2, 5, 25, and 100 milligrams.

SUMMARY:
This is an open-label study evaluating the efficacy and safety of lamotrigine (LTG) for the treatment of newly-diagnosed typical absence seizures. Subjects will be children and adolescents < 13 years of age. It will be conducted at multiple sites in the US. The study will consist of 4 phases: Screen Phase (up to 1 week), Baseline Phase (24 hours), Escalation Phase (up to 20 weeks) and Maintenance Phase (12 weeks). Subjects will receive increasing doses of LTG according to the dosing schedule until attaining seizure freedom as confirmed by hyperventilation (HV) for clinical signs and a 1-hr EEG at 2 consecutive weekly visits. At that point, subjects will move into the 12-week Maintenance Phase. Subjects who do not achieve seizure freedom upon reaching the maximum dose (10.2mg/kg/day) with the specified dose escalation will be discontinued from the study. During the Maintenance Phase, the investigators will use their best effort to maintain the subjects at the efficacious dose reached. If the subjects have unacceptable side effects or inadequate seizure control, the doses of study drug can be increased or decreased as specified in the dosing schedule. Safety will be assessed by monitoring adverse events, laboratory assessments, and serum lamotrigine levels. Health outcomes assessments will also be conducted.

ELIGIBILITY:
Inclusion criteria:

* Newly-diagnosed with absence epilepsy and never been treated with Anti-epileptic drugs (AEDs).
* Diagnosis demonstrated on one of two 5-minute hyperventilation tests.
* Investigator must judge that the subject and parent/guardian are likely to comply with all study procedures.
* Parent/guardian must given written informed consent. Subjects who are intellectually able to understand the concepts and procedures of the protocol must give assent by also signing the consent or by signing a separate assent form.
* Results of all screen assessments are judged to be clinically acceptable to the investigator and do not indicate any reasons why entry into the study would be contraindicated.

Exclusion criteria:

* Seizures are the result of a currently active, known, and identifiable intracerebral lesion.
* Has partial or generalized tonic-clonic seizures.
* Has a progressive neurological disorder defined as being unstable for at least 12 weeks prior to the Screen Phase.
* Has a psychiatric disorder requiring medication, or has had a past psychiatric condition that was both judged to be severe and required hospitalization.
* Has any clinically significant chronic cardiac, renal, or hepatic medical condition.
* Has a condition that affects the absorption, distribution, metabolism, or excretion of drugs.
* Is currently taking any psychoactive drugs to treat hyperactivity disorder or attention deficit disorder.
* Has taken any investigational drug within 12 weeks prior to the Screen Phase.
* Is sexually active.
* Is either pregnant (i.e., confirmed by pregnancy test at Screen) or breastfeeding.
* Has a clinically significant chronic medical disorder which the investigator and/or GSK medical monitor determine warrants exclusion.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2004-11-01 (Actual); Primary Completion 2006-04-22 (Actual); Study Completion 2006-04-22 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with no typical absence seizures for two consecutive weeks as confirmed by hyperventilation (HV) for clinical signs and 1-hour electroencephalogram (EEG) | Up to 8 months

SECONDARY OUTCOMES:
Freq of seizures pre/post-treatment with lamotrigine, proportion of subjects with >=25, 50 and 75% decrease in seizure frequency, proportion of subjects with >=25, 50 and 75% decrease in clinical signs. | Up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (22):
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Holmes GL, Frank LM, Sheth RD, Philbrook B, Wooten JD, Vuong A, Kerls S, Hammer AE, Messenheimer J. Lamotrigine monotherapy for newly diagnosed typical absence seizures in children. Epilepsy Res. 2008 Dec;82(2-3):124-32. doi: 10.1016/j.eplepsyres.2008.07.016. Epub 2008 Sep 7. PMID 18778916
- See also: Results for study LAM100118 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/LAM100118?search=study&study_ids=LAM100118#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: LAM100118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM100118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LAM100118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM100118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM100118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM100118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM100118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register